CLINICAL TRIAL: NCT01234753
Title: Follow up of Adults With Congenitally Malformed Hearts With Focus on Computer-Based Education and Psychosocial Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Ryhov County Hospital (Other); Kalmar County Hospital (Other); Skane University Hospital (Other)
Responsible Party: Helén Rönning, Department of Cardiology, Linköping University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SSKGUCH-1; M172-05 (Other: Regional Ethical Review Bords/Central Ethical Review Board)
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Last update posted 2010-11-04 (Estimated); Status verified 2009-01

CONDITIONS: Adults With Congenitally Malformed Hearts
Keywords: Adults with CHD; GUCH; Congenital heart disease; Computer-based education; Nursing
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Physicians

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- Usulal care (No Intervention): Usual care by a visit to physician at the hospital out-patient clinic
  Interventions: Other: Physician and nurse consultation

INTERVENTIONS:
Other: Physician and nurse consultation — Usual care by a visit to physician at the hospital out-patient clinic and computer-based and individual education and psychosocial support by a nurse-led session.

SUMMARY:
The number of adults with congenitally malformed hearts is increasing. According to a prospective population-based cohort study from Sweden (1992-2001) the prevalence of cardiovascular defects was 9.1 per 1,000 births, which is comparable to other presented prevalence data in the world.On the basis of 9 million inhabitants, Sweden should have approximately 82000 born with CHD and approximately 20000 will, in adult age, need regular follow up in cardiac care. This is a result of the greater improvements within paediatric heart surgery and there is an increasing demand for continuous follow up in the healthcare system.[2] Guidelines from the European Society of Cardiology and the Canadian Cardiovascular Society recommend follow-up oriented towards both medical and psychosocial problems.

Earlier studies have shown that adults with CHD have poor knowledge about their heart disease.The results are difficult to summarise because of the use of different instruments, methods and sample sizes. Most of the adults with CHD did not know their clinical diagnosis or what endocarditis was. However, we do not know if everyone in these studies was recommended endocarditis prophylactics or their definition of poor knowledge.

At present different programmes for adults with CHD are established in hospital outpatient clinics. These studies describe the established programmes. They also address the needs for development of care e.g. a multicenter approach, transitions from paediatric to adult health care, delivery care in Europe, programmes for pregnancy, how to provide clinical strategies, health care resource utilization or outpatient nursing clinic for adults with CHD. But there is a lack of knowledge regarding how education and psychosocial support should be given to adults with congenitally malformed hearts and what effects that can be achieved. The aim is to evaluate the effects of a nurse-led intervention consisting of education by a computer-based educational programme and psychosocial support to adults with congenitally malformed hearts.

DETAILED DESCRIPTION:
Sample: 114 adults with congenitally malformed hearts as ventricular septal defect, atrial septal defect, coarctation of the aortae, tetralogy of Fallot, complete transposition of the great arteries, congenitally corrected transposition of the great arteries, single ventricle, Ebstein anomaly, coarctation of the aortae, Eisenmenger syndrome and aortic valve stenosis.

Method and Measures: Randomised, controlled study where. the iIntervention-group will receive medical consultation, nurse consultation with psychosocial support, verbal and computer-based education. A care-plan with individual goals will be developed for each individual. Follow up of the care plan will be conducted after 1 month. The Control-group will receive: standard care with medical consultation.

Data will be collected at baseline and after 3 and 12 months. Instruments

* Knowledge instrument developed in Belgium , translated, further developed, tested in study 3. Now further reliability and validity tests in this study 4.
* Health related quality of life, Short Form 36 (SF-36). SF-36 has good validity and reliability and is adjust to Swedish circumstances • Anxiety and depression, Hospital Anxiety and Depression Scale, (HADS)
* General health related quality of life, Euroqol 5 dimensions (EQ-5D)
* Perceived control

ELIGIBILITY:
Inclusion Criteria:

* adults with uncomplicated congenitally malformed hearts (ventricular septal defect, atrial septal defect, coarctation of the aortae, aortic valve stenosis) and complicated congenitally malformed hearts (tetralogy of Fallot, complete transposition of the great arteries, congenitally corrected transposition of the great arteries, Ebstein anomaly and Eisenmenger syndrome),

Exclusion Criteria:

* complicating serious co-morbidity such as hereditary heart diseases (age-related coronary heart diseases, valve diseases), other diseases or life-threatening diseases, psychiatric illness or inability to read or understand Swedish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2006-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)